CLINICAL TRIAL: NCT04594811
Title: A Multicenter, Open-label, Phase 1 Dose Escalation ,Phase 2 Study of NT-I7 in Combination With Nivolumab in Subjects With Relapsed/Refractory Gastric or Gastro-Esophageal Junction or Esophageal Adenocarcinoma Who Progressed on or Intolerant to 2 or More Prior Lines of Systemic Therapy
Brief Title: NT-I7 in Combination With Nivolumab in Advanced Gastric, Gastro-Esophageal Junction or Esophageal Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company strategic decision
Sponsor: NeoImmuneTech (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIT-109; 2020-004175-41 (EudraCT Number)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-04

CONDITIONS: Gastric or Gastro-esophageal Junction (GEJ) or Esophageal Adenocarcinoma (EAC)
Keywords: NT-I7; Nivolumab; Dose escalation; Metastatic or Advanced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — efineptakin alfa; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): NT-I7 will be administered on Day 1 of alternate 4 weeks cycles (Cycle 1, 3, 5 etc.) (Q8W). Dosage will increase until the maximum tolerated dose (MTD) and/or the recommended phase 2 (RP2D) dose is reached.
  Nivolumab will be administered on Day 1 of every 4 week cycle (Q4W).
  Interventions: Drug: NT-I7; Drug: Nivolumab
- Phase 2: NT-I7 and Nivolumab (Experimental): NT-I7 will be administered on Day 1 of alternate 4 weeks cycles (Cycle 1, 3, 5 etc.) (Q8W) at the recommended phase 2 dose (RP2D) identified during Dose escalation phase.
  Nivolumab will be administered on Day 1 of every 4 week cycle (Q4W).
  Interventions: Drug: NT-I7; Drug: Nivolumab

INTERVENTIONS:
Drug: NT-I7 — Administered by intramuscular (IM) injection.
  Other Names: Efineptakin alfa; rhIL-7-hyFc
Drug: Nivolumab — Administered by intravenous (IV) injection.

SUMMARY:
The main purposes of the dose escalation part of this study is to determine the following in participants with gastric or gastro-esophageal junction (GEJ) or esophageal adenocarcinoma (EAC):

* Safety and tolerability of NT-I7 in combination with nivolumab
* Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RP2D)

The main purposes of Phase 2 of this study is to make a preliminary assessment of the antitumor activity and long-term survival of NT-I7 in combination with nivolumab in participants with gastric or GEJ or EAC.

Note, this trial was intended to be a Phase 1/2 trial (but the trial never moved forward to Phase 2).

ELIGIBILITY:
Inclusion Criteria:

1. Dose Escalation: Have histologically or cytologically confirmed locally advanced or metastatic solid tumor and can be either CPI-pretreated or CPI-naive.

   Phase 2: Have histologically or cytologically confirmed locally advanced or metastatic carcinoma of Gastric or Gastro-Esophageal Junction (GEJ) or Esophageal Adenocarcinoma (EAC) and who progressed on or intolerant to 2 or more prior lines of standard therapy including chemotherapy, immunotherapy, and targeted therapy.

   Note: GEJ adenocarcinomas are defined as tumors that have their center within 5 cm proximal and distal of the anatomical cardia, as described in the Siewert classification system (Siewert et al, 2000).
2. Have at least one measurable lesion according to RECIST 1.1.
3. Participants enrolling in the dose escalation phase may have biopsiable disease. Optional for participants to provide a) pre-treatment tumor tissue sample and b) on-treatment tumor biopsy.
4. At least 20 participants enrolled in the Phase 2 must agree to provide tumor tissue sample prior to the start of treatment.
5. Female participants are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks; if a female participant is of childbearing potential, she must agree to remain abstinent (refrain from heterosexual intercourse) or to follow instructions for one highly effective method of contraception for the duration of study treatment and for 5 months after the last dose of study treatment.
6. Non-sterile male participants who are sexually active with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or to follow instructions for one highly effective method of contraception for the duration of study treatment and for 3 months after the last dose of study treatment.

Exclusion Criteria:

1. Pregnant, or breastfeeding or expecting to conceive or father children within the study duration from screening through 5 months (for female participants) or 3 months (for male participants) after the last dose of study treatment.
2. Receiving chemotherapy or any anti-cancer therapy with half-life <1 week within 4 weeks or 5 half-lives, whichever is shorter, prior to first dose of study treatment.
3. Has received prior radiotherapy within 2 weeks of start of study treatment.
4. Has received treatment with complementary medications (excluding, herbal supplements, or traditional Chinese medications) to treat the disease under study within 2 weeks prior to the first dose of study treatment.
5. Subjects are eligible if CNS metastases are asymptomatic and do not require immediate treatment or have been treated and subjects have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment).
6. History of severe hypersensitivity reactions to monoclonal antibodies (mAbs) or intravenous immunoglobulin preparation.
7. Clinically significant cardiac disease.
8. Has a history of allergy or intolerance (unacceptable adverse events [AEs]) to study drug components or polysorbate-80-containing injections.

   Note: Polysorbate 80 is a buffer used to make NT-I7.
9. Has received a live vaccine within 4 weeks prior to the first dose of study drug. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed.
10. Has had an allogenic tissue/solid organ transplant or bone marrow transplant.
11. Subjects who were intolerable and discontinued from prior immune checkpoint inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Dose escalation: Number of participants who experience one or more treatment-emergent adverse events (TEAEs) | Up to 1 year
Dose escalation: Number of participants who experience one or more common terminology criteria for adverse events (CTCAE) grade ≥ 3 adverse events | Up to 1 year
Dose escalation: Number of participants who experience one or more dose limiting toxicities (DLTs) | Up to 1 year
Dose escalation: Number of participants who experience one or more common terminology criteria for adverse events (CTCAE) grade ≥ 3 dose limiting toxicities (DLTs) | Up to 1 year
Phase 2: Objective response rate (ORR) | Up to 2 years
  ORR is defined as the percentage of participants with a best overall response (BOR) of a complete response (CR) or partial response (PR), per RECIST 1.1.

SECONDARY OUTCOMES:
Duration of response (DoR) | Up to 3 years
  DOR is defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per RECIST 1.1.
Disease control rate (DCR) | Up to 3 years
  DCR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD), per RECIST 1.1.
Progression free survival (PFS) | Up to 3 years
  PFS is defined as the time from the first study treatment to the first occurrence of disease progression or death of any cause, whichever occurs first, per RECIST 1.1.
Phase 2: Overall survival (OS) | Up to 2 years
  OS is defined as the time from first study treatment to death from any cause.
Number of participants with anti-drug antibodies (ADA) to NT-I7 | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - The Center for Cancer & Blood Disorders, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Poland (2):
  - Centrum Medyczne Klara, Częstochowa
  - Pratia Poznań, Skorzewo